CLINICAL TRIAL: NCT00445081
Title: Prednisolone vs. Ciclosporine in Severe Atopic Eczema
Acronym: PROVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Jochen Schmitt, MD, MPH, Technical University Dresden
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUD_PROVE_001; EudraCT-Nr:2006-003667-31
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; prednisolone; ciclosporine; SCORAD; DLQI; QALY; WLQ
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Prednisolone
- 2 (Active Comparator)
  Interventions: Drug: Ciclosporine A

INTERVENTIONS:
Drug: Prednisolone
  Arms: 1
Drug: Ciclosporine A
  Arms: 2

SUMMARY:
To investigate the comparative efficacy of Ciclosporine A and Prednisolone in adult patients with severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients age >= 18 and < 55
* weight between 50 and 100 kg
* confirmed diagnosis of AE (UK working party criteria)
* objective SCORAD > 40
* DLQI > 10
* resistancy against topical treatment options including steroids and calcineurin-inhibitors

Exclusion Criteria:

* participation to another clinical trial within the last 4 weeks before baseline
* pregnant or breastfeeding
* women of childbearing potential without adequate contraception
* allergy against prednisolone or Ciclosporine A
* acute bacterial or viral infection
* malignant tumor in personal history
* diabetes mellitus
* arterial hypertension
* Glaucoma
* peptic ulcer
* severe osteoporosis
* tuberculosis in personal history
* colitis ulcerosa
* diverticulitis
* concurrent treatment with chloroquin, Mefloquin, Statins, Warafin
* Creatinin Clearance < 60 ml /min
* UV treatment within 8 weeks before inclusion
* ongoing systemic immunosuppressive treatment
* planned vaccination within 8 weeks before study entry, during study and 2 weeks after end of study
* Poliomyelitis
* Lymphadenitis after BCG vaccination
* Hyperuricaemia
* chronic liver disease
* Xeroderma pigmentosum, Cockaye-Syndrome, Bloom Syndrome
* Psychiatric co-morbidity
* drug or alcohol abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2007-03; Primary Completion 2009-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
stable remission in both treatment groups

SECONDARY OUTCOMES:
response rate in both treatment groups
relapse rate in both treatment groups
mean change in objective SCORAD in both treatment groups
mean change in HRQL (DLQI) in both treatment groups
change in disease symptoms (POEM)in both treatment groups
Cost-effectiveness of both treatments
Tolerability and Safety
change in presenteeism in both treatment groups
patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Jochen M Schmitt, MD MPH, Principal Investigator — Dpt. of Dermatology, TU Dresden, Fetscherstr 74, D-01307 Dresden
Locations (5):
- University Hospital of Dermatology and Venerology Graz, Graz, Austria
- Germany (4):
  - Dept. of Dermatology, Medical Faculty, TU Dresden, Dresden
  - Dpt. of Dermatology, Medical Faculty Eppendorf, Hamburg
  - University Hospital Kiel, Kiel
  - Dpt. of Dermatology, University Hospital Münster, Münster

REFERENCES:
- [Derived] Schmitt J, Schakel K, Folster-Holst R, Bauer A, Oertel R, Augustin M, Aberer W, Luger T, Meurer M. Prednisolone vs. ciclosporin for severe adult eczema. An investigator-initiated double-blind placebo-controlled multicentre trial. Br J Dermatol. 2010 Mar;162(3):661-8. doi: 10.1111/j.1365-2133.2009.09561.x. Epub 2009 Oct 26. PMID 19863501